CLINICAL TRIAL: NCT01487525
Title: Assessment of Efficacy of Low Intensity Resistance Training in Men at Risk for Symptomatic Knee Osteoarthritis
Acronym: PBFR3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Neil A Segal, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 201109738-MOD
Record Dates: First submitted 2011-12-01; First posted 2011-12-07 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Knee Osteoarthritis
Keywords: symptomatic knee osteoarthritis; partial blood flow restriction; knee extensor strength
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBFR- (Placebo Comparator): double leg press without application of partial blood flow restriction to the upper leg
  Interventions: Other: Double leg press without partial blood flow restriction
- PBFR+ (Experimental): double leg press with application of partial blood flow restriction to the upper leg
  Interventions: Device: Double leg press with partial blood flow restriction

INTERVENTIONS:
Device: Double leg press with partial blood flow restriction — double isotonic and isokinetic leg press extension with application of partial blood flow restriction to the upper leg
  Arms: PBFR+
Other: Double leg press without partial blood flow restriction — double isotonic and isokinetic leg press extension without application of partial blood flow restriction to the upper leg
  Arms: PBFR-

SUMMARY:
The purpose of this research study is to determine whether low intensity resistance training with concurrent application of a peripheral blood flow restriction device to the exercising limb will elicit increased quadriceps strength, functional gains, ability to complete knee-related activities of daily living, mobility, and quality of life in individuals at risk for developing symptomatic knee osteoarthritis (OA). It is known that higher quadriceps strength is protective against developing symptomatic knee OA.1 However, people at risk for knee OA frequently do not tolerate the high intensity resistance training that is generally believed necessary to increase muscle strength. Partial blood flow restriction (PBFR) to the exercising muscle has been reported to result in strength gains, while requiring lower levels of joint loading.2 This method may be better tolerated, enabling efficacious exercise in older adults who may not tolerate high knee joint loads.

To asses the efficacy of a 4 week low-intensity resistance training program with concurrent application of PBFR to the exercising limbs to improve quadriceps strength and size, leg muscle power, and mobility in individuals at risk for developing symptomatic knee osteoarthritis,we will test the following hypotheses. In comparison with low-intensity resistance training without use of PBFR, a four-week low-intensity resistance-training program with PBFR will:

Primary Hypothesis: Increase (a) double leg-press 1RM strength and (b) isokinetic knee extensor strength

Secondary Hypotheses:

1. Increase quadriceps muscle volume assessed by MRI
2. Increase lower limb muscle power on (a) double leg-press at 40% 1RM and (b) a timed stair climb
3. Not adversely effect knee pain or quality of life assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire

DETAILED DESCRIPTION:
Over 9.3 million adults over the age of 60 are afflicted with symptomatic knee osteoarthritis (OA) characterized by radiographic findings and consistent knee pain or stiffness. Furthermore, our research has indicated that reduced strength is a risk factor for incident symptomatic knee OA and progressive knee OA in women.1, 3 In light of this finding, there is a need to increase quadriceps strength to attenuate worsening of this disease. Studies and practice have long indicated that high intensity resistance training is the most efficient means of eliciting skeletal muscle hypertrophy and strength gains.2, 4 The American College of Sports Medicine as well as the National Strength and Conditioning Association have indicated that a resistance training intensity of greater than 65% of the one-repetition maximum (1 RM) is the minimum intensity needed to achieve desired muscle hypertrophy and strength gains.2, 4 This is problematic for those suffering from symptomatic knee OA. Loading an already painful joint at 65% of (1 RM) would be poorly tolerated and possibly injurious for an individual already suffering knee pain and stiffness during activities of daily living. With the inability to perform the exercises prescribed to elicit the necessary strength gains, knee OA sufferers find themselves unable to alleviate debilitating pain that can result in significant decreases in quality of life. Fortunately, a method of training, called partial blood flow restriction (PBFR), may offer older adults and particularly those with knee OA, the ability to develop the strength gains necessary to attenuate disease progression without requiring deleterious joint loading. There is mounting evidence that this training modality serves as a stimulator of muscle growth even when performed at relatively low intensities.

PBFR was developed in Japan. Its basic principles involve the restriction of blood flow to the exercising muscle with the purpose of increasing muscle mass. However, participants are able to elicit similar strength gains performing exercises at, for example, only 30% of 1RM to those attained through conventional high intensity resistance training. Current PBFR training methods are the result of 40 years of research and development.5 Recent studies have demonstrated efficacy and some mechanisms for the effect of PBFR training eliciting significant isometric and isokinetic strength gains as well as increasing ability of adults to perform functional tasks.6 Exercising at only 30% 1RM, PBFR training may benefit older adults suffering from knee OA by enabling development of the strength necessary to protect against disease worsening while avoiding the need to load the joint at deleterious levels.

This study is a follow-up study to IRB#201101711 that we completed earlier this year. That study demonstrated tolerance and safety of the protocol. However, the increases in strength were of a smaller magnitude than we hoped to elicit. The protocol for this follow-up study is very similar to the prior study. We have made some changes in an effort to maintain tolerability and safety, while hopefully eliciting a greater clinical benefit. Specifically, we have reduced the study duration from 9 to 4 weeks and have selected a more efficient exercise protocol that will both reduce subject burden while also halving the length of time that the PBFR cuffs will be worn for each exercise session. The prior study was too gentle to strengthen the quadriceps muscles, so we have increased the resistance from 15% of their maximum to 30% of their maximum. This is still low intensity compared with usual weight lifting that would be at >65%. We believe that these changes will increase benefit to participants while reducing the time burden.

Literature cited

1. Segal NA, Torner JC, Felson D, Niu J, Sharma L, Lewis CE et al. Effect of thigh strength on incident radiographic and symptomatic knee osteoarthritis in a longitudinal cohort. Arthritis Rheum 2009;61(9):1210-7.
2. Abe T, Kearns CF, Sato Y. Muscle size and strength are increased following walk training with restricted venous blood flow from the leg muscle, Kaatsu-walk training. J Appl Physiol 2006;100(5):1460-6.
3. Segal NA, Glass NA, Torner J, Yang M, Felson DT, Sharma L et al. Quadriceps weakness predicts risk for knee joint space narrowing in women in the MOST cohort. Osteoarthritis Cartilage 2010;18(6):769-75.
4. Abe T, Kearns CF, Manso Filho HC, Sato Y, McKeever KH. Muscle, tendon, and somatotropin responses to the restriction of muscle blood flow induced by KAATSU-walk training. Equine Vet J Suppl 2006(36):345-8.
5. Sato Y. The history and future of KAATSU Training. Int J KAATSU Training Research 2005;1:1-5.
6. Fry CS, Glynn EL, Drummond MJ, Timmerman KL, Fujita S, Abe T et al. Blood flow restriction exercise stimulates mTORC1 signaling and muscle protein synthesis in older men. J Appl Physiol;108(5):1199-209.
7. Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc 2000;32(12):2035-9.
8. Takano H, Morita T, Iida H, Asada K, Kato M, Uno K et al. Hemodynamic and hormonal responses to a short-term low-intensity resistance exercise with the reduction of muscle blood flow. Eur J Appl Physiol 2005;95(1):65-73.
9. Fujita S, Abe T, Drummond MJ, Cadenas JG, Dreyer HC, Sato Y et al. Blood flow restriction during low-intensity resistance exercise increases S6K1 phosphorylation and muscle protein synthesis. J Appl Physiol 2007;103(3):903-10.
10. Iida H, Kurano M, Takano H, Kubota N, Morita T, Meguro K et al. Hemodynamic and neurohumoral responses to the restriction of femoral blood flow by KAATSU in healthy subjects. Eur J Appl Physiol 2007;100(3):275-85.
11. Cook SB, Clark RC, Ploutz-Snyder LL. Effects of Exercise Load and Blood-Flow Restriction on Skeletal Muscle Function. Med Sci Sports Exerc 2007.

ELIGIBILITY:
Inclusion Criteria:

* male
* ≥ 45 years
* has at least one of the following: BMI≥25, frequent knee symptoms on most of the last 30 days, history of knee injury which rendered individual unable to walk without assistance for at least 2 days, history of knee surgery, diagnosis of knee osteoarthritis

Exclusion Criteria:

* Resistance training at any time in the last 3 months prior to study
* Bilateral knee replacement
* Lower limb amputation
* Lower limb surgery in the last 6 months that affects walking ability or ability to exercise
* Back, hip or knee problems that affect walking ability or ability to exercise
* Unable to walk without a cane or walker
* Inflammatory joint or muscle disease such as rheumatoid or psoriatic arthritis or polymyalgia rheumatica
* Multiple sclerosis
* Known neuropathy
* Self-report of Diabetes
* Currently being treated for cancer or having untreated cancer
* Terminal illness (cannot be cured or adequately treated and there is a reasonable expectation of death in the near future)
* Peripheral Vascular Disease
* History of myocardial infarction or stroke in the last year
* History of deep venous thrombosis
* Chest pain during exercise or at rest
* Use of supplemental oxygen
* Inability to follow protocol (e.g. lack of ability to attend visits or understand instructions)
* Staff concern for subject health (such as history of dizziness/faintness or current restrictions on activity)
* Concurrent study participation
* Unable to attend more than 2 days within any 1 week or unable to attend 4 or more sessions during the study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 subjects were enrolled. Prior to starting the study, 2 participants dropped out due to lack of time. Since they discontinued after consent, but prior to any measurements or interventions, no data is available for these 2. Data is available for the 42 subjects who started the study.
Groups:
- PBFR-: strength training exercise without partial blood flow restriction
  double leg press without partial blood flow restriction: double leg press extension without application of partial blood flow restriction to the upper leg
- PBFR+: strength training exercise with partial blood flow restriction
  double leg press with partial blood flow restriction: double leg press extension with application of partial blood flow restriction to the upper leg
Period: Overall Study
Arm/Group | PBFR- | PBFR+
Started | 22 | 20
Completed | 22 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Control BFR p-value Age (years) 56.1±7.7 58.4±8.7 0.377
Groups:
- Total: Total of all reporting groups
Arm/Group | PBFR- | PBFR+ | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (7.7) | 58.4 (8.7) | 57.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 20 | 42
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Isotonic Leg Press 1RM
Description: double leg press 1 rep maximum strength
Time Frame: 0,6 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PBFR- | PBFR+
Number analyzed (Participants) | 22 | 19
percent change | 4.7 (1.3) | 3.1 (0.9)

2. Secondary Outcome: Isokinetic Knee Extensor Strength
Time Frame: 0, 6 weeks
Measure: Mean (Standard Error); unit: percent change
Arm/Group | PBFR- | PBFR+
Number analyzed (Participants) | 22 | 19
percent change | 6.7 (2.3) | 0.4 (2.4)

3. Secondary Outcome: Knee Pain
Description: Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire Pain Sub-Scale (0-100); larger absolute values represent less pain; a positive % changes indicates a reduction in pain
Time Frame: 0, 6 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | PBFR- | PBFR+
Number analyzed (Participants) | 22 | 19
Percent change | 14.2 (7.2) | 4.9 (3.3)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | PBFR- | PBFR+
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No